CLINICAL TRIAL: NCT06817954
Title: A Prospective, Single-center, Double-arm Clinical Study to Evaluate the Effectiveness and Safety of Mastectomy Combined With Immediate Breast Reconstruction in Breast Cancer
Brief Title: To Evaluate the Effectiveness and Safety of Mastectomy Combined With Immediate Breast Reconstruction in Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-MCWIBR-20250205
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Endoscopic-assisted mastectomy and immediate breast reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic-assisted mastectomy and immediate breast reconstruction (Experimental): endoscopic-assisted mastectomy and immediate breast reconstruction
  Interventions: Procedure: endoscopic-assisted mastectomy and immediate breast reconstruction
- mastectomy and immediate breast reconstruction (Experimental): mastectomy and immediate breast reconstruction
  Interventions: Procedure: mastectomy and immediate breast reconstruction

INTERVENTIONS:
Procedure: endoscopic-assisted mastectomy and immediate breast reconstruction — endoscopic-assisted mastectomy and sentinel lymph node biopsy/axillary lymph node dissection in the management of breast cancer
  Arms: endoscopic-assisted mastectomy and immediate breast reconstruction
Procedure: mastectomy and immediate breast reconstruction — conventional mastectomy and sentinel lymph node biopsy/axillary lymph node dissection in the management of breast cancer
  Arms: mastectomy and immediate breast reconstruction

SUMMARY:
The new technology of endoscopic-assisted system, as an emerging technology, has shown certain application prospects in breast surgery. However, the new technology of endoscopic-assisted mastectomy and immediate breast reconstruction in China in the treatment of breast cancer is still in the exploratory stage and needs to be further improved. This prospective, single-center, double-arm clinical study was conducted to use the endoscopic-assisted system and evaluate the effectiveness and safety of the mastectomy combined with immediate breast reconstruction in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, aged 18-75 years old; The pregnancy test (-) and reliable contraceptive methods are required for premenopausal and perimenopausal patients;
2. Patients with the diagnosed breast cancer confirmed by core needle biopsy and unilateral operation was performed; Breast cancer patients with tumor node metastasis stage 0-III according to the 8th edition of the American Joint Commission on Cancer; Preoperative clinical examination or imaging evaluation shows that the distance between the tumor and the Nipple Areolar Complex (NAC) is more than 1cm. The tumor has a diameter of 2-3 cm and can be located in any quadrant or reduced to 3 cm through preoperative neoadjuvant chemotherapy. The distance between the lesion and the skin should be at least 8-10 mm;
3. There is no clinical or imaging evidence to prove that the tumor has invaded the skin, chest wall, or nipple areola complex;
4. There are indications for breast preservation, but the patient has a strong desire for reconstruction and is unwilling to undergo breast preservation surgery;
5. Preventive mastectomy (BRCA1/2 malignant mutation with obvious family history of breast cancer and other high-risk groups);
6. Preoperative clinical manifestations and imaging data showed no distant metastasis;
7. No history of breast cancer or other serious underlying diseases in the past;
8. Karnofsky performance status score ≥ 70;
9. Eastern Cooperative Oncology Group score ≤ 2 ;
10. The surgical procedure includes endoscopic-assisted/conventional mastectomy, sentinel lymph node biopsy/axillary lymph node dissection and immediate breast reconstruction;
11. Participants are able to understand the research process, voluntarily join the study, sign informed consent forms, have good compliance, and cooperate with follow-up;
12. No swallowing difficulties; No shoulder joint movement disorders;
13. Complete clinical data.

Exclusion Criteria:

1. Male breast cancer or inflammatory breast cancer;
2. Metastatic breast cancer (stage IV); Tumor invasion of the skin, pectoralis major muscle, or NAC;
3. The clinical data is basically incomplete;
4. Previously received chemotherapy in an external hospital or has undergone tumor resection in an external hospital;
5. Bilateral breast cancer surgery;
6. Other surgical methods;
7. Preoperative distant metastasis or supraclavicular lymph node dissection;
8. Complicated with other malignant tumors or had malignant tumors other than breast cancer in recent 5 years;
9. The serious disease of non malignant tumors combined will affect the patient's compliance or put the patient in a dangerous state;
10. Dementia, intellectual disability, or any mental illness that hinders understanding of informed consent forms.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival rate | Ten years
  Local recurrence refers to the recurrence of the chest wall or breast on the same side as the surgical site.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No